CLINICAL TRIAL: NCT06301113
Title: The Antimicrobial Impact of CBD-infused Lozenges on Streptococcus Mutans When Compared to Sugar Free Candy, on Thirty Adults Who Meet the Inclusion Criteria, Randomly Placed Into Two Groups Utilizing Quantitative Polymerized Chain Reaction Bacterial Analysis Technique.
Brief Title: This Research Study Examines the Effects of Cannabidiol-infused Candy on Reducing the Bacteria Causing Tooth Decay, When Comparing it to a Sugar Free Candy on Adults.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Coast University (Other)
Responsible Party: Principal Investigator, Jila Torabi, Assistant Professor, West Coast University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: IRB#: 01202023_torabiDH_CBDloz
Record Dates: First submitted 2024-03-01; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Tooth Decay
Keywords: CBD, streptococcus mutans
MeSH Terms: conditions — Dental Caries; Color Vision Defects

STUDY DESIGN:
Intervention Model Description: 30 Participants were randomly assigned to groups A (experimental group)and B (Control group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 300 Nano mg CBD Candy (Experimental)
  Interventions: Dietary Supplement: CBD infused candy
- Sugar free raspberry flavor candy (Placebo Comparator)
  Interventions: Dietary Supplement: Sugar free Candy

INTERVENTIONS:
Dietary Supplement: CBD infused candy — 300 Nano mg CBD Candy cherry flavor
  Arms: 300 Nano mg CBD Candy
Dietary Supplement: Sugar free Candy — Raspberry flavored sugar free candy
  Arms: Sugar free raspberry flavor candy

SUMMARY:
The goal of this clinical trial is to compare the effect of CBD candy versus sugar free candy on reducing the number of bacteria causing tooth decay, in adults The main question is to see whether CBD have any effect on reducing the number of Streptococcus mutans, in the oral cavity the main bacteria causing tooth decay.

Participants will be randomly placed in a group, and assigned to take either CBD-infused lozenge (if in the experimental group) or a sugar-free candy (if in the control group) once a day for 15 days.

A sample of saliva will be collected and analyzed in a lab before and after consumption of the candy to see whether either product could reduce the harmful bacteria in the mouth.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 years or older, that were not taking any antibiotics, using prescribed toothpaste or mouthwash, who were not experiencing any tooth ache or mouth sores, have not visited the dentist within the past 48 hours, who willingly signed a consent form agreed to participate and be available on specific dates set by investigators and followed the recommended regimen for 15 days were included in the study. The suggested regimen involved consuming one candy in the evening at approximately the same time, allowing it to dissolve in the mouth without crushing it. Furthermore, individuals who could abstain from alcohol consumption for at least 12 hours before saliva collection on day 1 and day 15 and refrain from food or drink (except water) for preferably 2 hours were also eligible to participate in this clinical trial.

Exclusion Criteria:

Encompassed individuals taking or recently completing an antibiotic regimen within two weeks before participation. Participants with allergies to specific substances, such as propriety broad spectrum nano hemp extract, isomalt, organic stevia, natural or artificial cherry flavoring, natural coloring, maltitol syrup, or citric acid, were also excluded. Further exclusion criteria included participants using professional-strength anti-cavity or anti-gingivitis products, individuals experiencing toothache or mouth sores, and those who had visited a dentist within the last 48 hours. In addition, participants who did not meet the saliva collection guideline protocols were excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-02-11 (Actual); Study Completion 2023-02-11 (Actual)

PRIMARY OUTCOMES:
To investigate the impact of CBD-infused lozenges on Streptococcus mutans, by employing quantitative polymerase chain reaction (qPCR) for bacterial analysis. | 15 days
  Align with the purpose of this clinical trial was to investigate the effect of CBD-infused lozenges on S. mutant, this clinical trial considered the dependent variable to be S. mutans gene expression as well as the 16S rRNA sequence, which is the universal gene in all bacteria measured in a continuous qPCR amplification cycle. The changes in the relative abundance of S. mutans pre and post-CBD lozenge consumption for 15 days were compared with the sugar-free candy and were measured via qPCR laboratory analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- West Coast University, Anaheim, California, United States

IPD SHARING:
Plan to Share IPD: No